CLINICAL TRIAL: NCT03875144
Title: Phase II Multicenter Randomized Trial Evaluating the Association of PIPAC and Systemic Chemotherapy Versus Systemic Chemotherapy Alone as 1st-line Treatment of Malignant Peritoneal Mesothelioma
Brief Title: Treatment of Malignant Peritoneal Mesothelioma (MESOTIP)
Acronym: MESOTIP
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: This decision was taken following the occurrence of three cases of serious and unexpected suspected adverse reactions (SUSARs), specifically febrile neutropenia, in participants assigned to the experimental arm combining PIPAC with systemic chemothe
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2019-03 MES
Record Dates: First submitted 2019-03-04; First posted 2019-03-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Peritoneal Mesothelioma; Peritoneal Carcinomatosis
Keywords: Peritoneal mesothelioma; PIPAC; Surgical oncology; Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Cisplatin; Doxorubicin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- association of PIPAC and systemic chemotherapy (Experimental): 4 PIPAC of Cisplatin 10.5mg/m² + Doxorubicin 2.1 mg/m² every 6 weeks alternating with standard intravenous chemotherapy for mesothelioma (Cisplatin 75mg/m² + Pemetrexed 500mg/m²)
  Interventions: Procedure: PIPAC; Drug: Cisplatin; Drug: Pemetrexed
- systemic chemotherapy alone (Active Comparator): 6 cycles of Cisplatin 75mg/m² + Pemetrexed 500mg/m²
  Interventions: Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Procedure: PIPAC — Pressurized IntraPeritoneal Aerosol Chemotherapy of Cisplatin 10.5mg/m² + Doxorubicin 2.1 mg/m² every 6 weeks
  Other Names: Cisplatin; Doxorubicin
  Arms: association of PIPAC and systemic chemotherapy
Drug: Cisplatin — standard intravenous chemotherapy for mesothelioma (Cisplatin 75mg/m² + Pemetrexed 500mg/m²)
Drug: Pemetrexed — standard intravenous chemotherapy for mesothelioma (Cisplatin 75mg/m² + Pemetrexed 500mg/m²)

SUMMARY:
MESOTIP is a randomized trial evaluating the association of PIPAC and systemic chemotherapy versus systemic chemotherapy alone as 1st-line treatment of Malignant Peritoneal Mesothelioma In this study, patients in the experimental arm will be treated by 4 PIPAC (Cisplatine+Doxorubicine) alternating with 6 cycles of standard intravenous chemotherapy (Cisplatine+Pemetrexed).

MESOTIP aim to show an improvement of the overall survival in the experimental arm.

DETAILED DESCRIPTION:
Malignant peritoneal mesothelioma (MPM) is a rare tumoral disease characterized by the diffuse involvement of the peritoneal serosa. The incidence of all mesotheliomas is estimated quite differently in various reports with the highest rates in industrialized countries. In France, the estimated incidence is 300 cases/year. Three types of malignant mesotheliomas are described in the WHO classification: epithelioid, sarcomatoid and biphasic.

The standard treatment of MPM is surgery. It has been shown that cytoreductive surgery (CRS) associated to hyperthermic intraperitoneal chemotherapy (HIPEC) improves prognosis resulting in a median overall survival of 29.5 months to 53 months and an 5 years overall survival rate ranging between 39 to 63%. Cytoreductive surgery should be complete or almost complete (CCR0/1) as macroscopic residual disease deteriorates prognosis.

However some patients are not eligible for surgery due to the locoregional extension of the disease. Although debulking surgery may still be considered, its results are less encouraging than CRS and HIPEC.

The neoadjuvant treatment combining Cisplatin and Pemetrexed became a routinely applied option for initially unresectable patients after the publication of an open-label study inspired by previous results of a randomized trial in pleural mesothelioma. This study showed a benefit in median survival of 5 months and an increase in the response rate of 10%. Ever since, other phase II studies were proposed but their benefit is still limited. Pleural mesothelioma which is more common and represents the model of choice for the treatment of peritoneal mesothelioma has also benefitted from phase III studies analyzing the addition of a targeted therapy (Bevacizumab) and phase II trials proposing immunotherapy.

By contrast, peritoneal mesothelioma was the setting of choice for testing intraperitoneal administration of chemotherapy either as early postoperative intraperitoneal chemotherapy (EPIC) or as neoadjuvant intraperitoneal chemotherapy. Both studies offered promising results showing a sensitivity of MPM to intraperitoneal administration.

Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) has recently been developed and shows interesting results in the neoadjuvant context of several peritoneal carcinomatoses while producing little toxicity. PIPAC is a modality of repeated administration of intraperitoneal chemotherapy during laparoscopy using aerosols at the pressure of the capnoperitoneum (12mmHg). Data from ex-vivo, in-vivo and human studies demonstrated a higher local drug bioavailability when compared to liquid IP chemotherapy. PIPAC was tested in the setting of malignant mesothelioma showing encouraging results.

In our study MESOTIP, patients in the experimental arm will be treated by 4 PIPAC (Cisplatine+Doxorubicine) alternating with 6 cycles of standard intravenous chemotherapy (Cisplatine+Pemetrexed).

Although retrospective reports showing the interest of PIPAC in the neoadjuvant setting for different peritoneal carcinomatosis origins were published, MESOTIP would be the first study to combine PIPAC to systemic chemotherapy in the first-line of treatment and to only include patients not eligible for surgical treatment and proposing a complete cytoreductive surgery associated to HIPEC for patients converted to resectability.

MESOTIP aim to show an improvement of the overall survival in the experimental arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. PS (or WHO) <2
3. Histologically-confirmed diagnosis of peritoneal malignant mesothelioma
4. No previous line of treatment (both medical and surgical oncologic treatments) for this disease
5. Peritoneal Carcinomatosis Index (PCI)>27 or at least 4 on the small bowel with serosal involvement contraindicating the cytoreductive surgery because of the impossibility to preserve a length >=1.5 m of uninvolved small bowel
6. Written and dated informed consent
7. Affiliated to the French national social security system

Exclusion Criteria:

1. WHO performance status ≥ 2
2. Any contraindication to chemotherapy and/or radiotherapy
3. Any contraindication to repeated laparoscopy
4. Symptomatic cardiac or coronary insufficiency
5. Severe renal insufficiency
6. Progressive active infection or any other severe medical condition
7. Intestinal occlusion non responsive to medical treatment
8. Other cancer treated within the last 2 years except in situ cervical carcinoma or basocellular/spinocellular carcinoma
9. Pregnant or breast-feeding woman
10. Previously operated patients where laparoscopy is not feasible
11. Persons deprived of liberty or under guardianship or incapable of giving consent
12. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
overall survival | from randomization of first patient until the database cut-off
  The overall survival is defined as the time from the date of randomization to the date of death from any cause

SECONDARY OUTCOMES:
Response to treatment using PFS | week 10, week21,every 4 months during 2 years
  Progression free survival (PFS) defined as the time from the date of randomization to the date of any progression or death. PFS will be described with median PFS, 1 and 2y-PFS rate
Adverse event | during treatment
  Safety according to CTCAE v5.0. Complications related to PIPAC will also be defined according to CTCAE v5.0 as recent publications in the field of peritoneal carcinomatosis suggest that this classification is more reliable when compared with the Clavien Dindo classification for the peritoneal carcinomatosis surgery
Feasibility of compliance | Week 21
  Feasibility rate of compliance defined as the percentage of patients who received 6 cycles of systemic chemotherapy and 4 PIPAC (for experimental arm).
Conversion to resectability | surgery
  Conversion to resectability rate defined as the percentage of patients eligible for cytoreductive surgery and HIPEC at the end of the treatment out of the total number of patients. Patients are eligible for surgery if preservation of at least 1.5 m of small bowel and of at least 2 m of lower gastrointestinal tube is feasible in case of complete cytoreduction.
Quality of life evaluation | baseline, week10, week21, FU every 4 months during 2 years
  Quality of life EORTC QLQ-C30 questionnaires according to EORTC Guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Olivia SGARBURA, MD, Principal Investigator — Institut régional du Cancer de Montpellier
Locations (1):
- Institut réginal du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim J, Bhagwandin S, Labow DM. Malignant peritoneal mesothelioma: a review. Ann Transl Med. 2017 Jun;5(11):236. doi: 10.21037/atm.2017.03.96. PMID 28706904
- [Background] Boffetta P. Epidemiology of peritoneal mesothelioma: a review. Ann Oncol. 2007 Jun;18(6):985-90. doi: 10.1093/annonc/mdl345. Epub 2006 Oct 9. PMID 17030547
- [Background] Bossard N, Velten M, Remontet L, Belot A, Maarouf N, Bouvier AM, Guizard AV, Tretarre B, Launoy G, Colonna M, Danzon A, Molinie F, Troussard X, Bourdon-Raverdy N, Carli PM, Jaffre A, Bessaguet C, Sauleau E, Schvartz C, Arveux P, Maynadie M, Grosclaude P, Esteve J, Faivre J. Survival of cancer patients in France: a population-based study from The Association of the French Cancer Registries (FRANCIM). Eur J Cancer. 2007 Jan;43(1):149-60. doi: 10.1016/j.ejca.2006.07.021. Epub 2006 Nov 3. PMID 17084622
- [Background] Alexander HR Jr, Li CY, Kennedy TJ. Current Management and Future Opportunities for Peritoneal Metastases: Peritoneal Mesothelioma. Ann Surg Oncol. 2018 Aug;25(8):2159-2164. doi: 10.1245/s10434-018-6337-5. Epub 2018 Feb 8. PMID 29423664
- [Background] Yan TD, Deraco M, Baratti D, Kusamura S, Elias D, Glehen O, Gilly FN, Levine EA, Shen P, Mohamed F, Moran BJ, Morris DL, Chua TC, Piso P, Sugarbaker PH. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy for malignant peritoneal mesothelioma: multi-institutional experience. J Clin Oncol. 2009 Dec 20;27(36):6237-42. doi: 10.1200/JCO.2009.23.9640. Epub 2009 Nov 16. PMID 19917862
- [Background] Baratti D, Kusamura S, Cabras AD, Bertulli R, Hutanu I, Deraco M. Diffuse malignant peritoneal mesothelioma: long-term survival with complete cytoreductive surgery followed by hyperthermic intraperitoneal chemotherapy (HIPEC). Eur J Cancer. 2013 Oct;49(15):3140-8. doi: 10.1016/j.ejca.2013.05.027. Epub 2013 Jul 4. PMID 23831335
- [Background] Helm JH, Miura JT, Glenn JA, Marcus RK, Larrieux G, Jayakrishnan TT, Donahue AE, Gamblin TC, Turaga KK, Johnston FM. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy for malignant peritoneal mesothelioma: a systematic review and meta-analysis. Ann Surg Oncol. 2015 May;22(5):1686-93. doi: 10.1245/s10434-014-3978-x. Epub 2014 Aug 15. PMID 25124472